CLINICAL TRIAL: NCT06703177
Title: Phase IB/II Study of Safety, Tolerability and Efficacy of SHR-1826 for Injection in Combination With Other Antitumor Therapies in Subjects With Solid Tumors
Brief Title: A Study of SHR-1826 for Injection in Combination With Other Antitumor Therapies in Subjects With Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1826-201
Record Dates: First submitted 2024-11-19; First posted 2024-11-25 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Bevacizumab; Fluorouracil; Leucovorin; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single group (Experimental)
  Interventions: Drug: SHR-1826; Drug: SHR-4642; Drug: SHR-9839; Drug: SHR-8068; Drug: Bevacizumab Injection; Drug: Fluorouracil Injection; Drug: Calcium Folinate Injection; Drug: Adebrelimab Injection; Drug: Capecitabine tablets

INTERVENTIONS:
Drug: SHR-1826 — SHR-1826
Drug: SHR-4642 — SHR-4642
Drug: SHR-9839 — SHR-9839
Drug: SHR-8068 — SHR-8068
Drug: Bevacizumab Injection — Bevacizumab Injection
Drug: Fluorouracil Injection — Fluorouracil Injection
Drug: Calcium Folinate Injection — Calcium Folinate Injection
Drug: Adebrelimab Injection — Adebrelimab Injection
Drug: Capecitabine tablets — Capecitabine tablets, oral.

SUMMARY:
This is an open label, multi-center, multiple dose Phase IB/II study to evaluate the safety, tolerability and efficacy of SHR-1826 for injection in subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation and written informed consent;
2. 18-75 years older, no gender limitation;
3. Eastern Cooperative Oncology Group (ECOG) score: 0-1;
4. With a life expectancy ≥ 3 months;
5. Pathologically diagnosed advanced solid tumor;
6. Be able to provide fresh or archived tumour tissue;
7. At least one measurable lesion according to RECIST v1.1;
8. Adequate bone marrow reserve and organ function;
9. Contraception is required during clinical trials, and pregnancy tests must be negative for women of childbearing age within 7 days before the first dose.

Exclusion Criteria:

1. Meningeal metastasis history or clinical symptoms of central nervous system metastasis;
2. Previous or co-existing malignancies;
3. Spinal cord compression that was not treated radically by surgery and/or radiotherapy was excluded;
4. Uncontrollable tumor-related pain;
5. Previously received antiboy-coupled drug therapy with topoisomerase I inhibitor toxin; Previously received EGFR/c-Met double antibody;
6. Received systemic antitumor therapy before the first dose;
7. Have undergone major surgery other than diagnosis or biopsy within 28 days prior to initial dosing; Minor traumatic surgery within 7 days prior to first dosing;
8. For the first time, a study was conducted to treat patients with radiation therapy exceeding the prescribed dose before study treatment;
9. Received Other investigational drugs treatments 4 weeks prior to the initiation of the study treatment;
10. Unresolved CTCAE 5.0>grade 2 toxicities from previous anticancer therapy;
11. A history of interstitial pneumonia/non-infectious pneumonia;
12. Accompanied by uncontrolled pleural effusion and pericardial effusion; Moderate or severe ascites with clinical symptoms;
13. Study the presence of intestinal obstruction or the presence of signs or symptoms of intestinal obstruction 6 months before first dosing;
14. With poorly controlled or severe cardiovascular disease;
15. Active hepatitis B, hepatitis C;
16. Patients with a history of immunodeficiency;
17. Severe infection 30 days before the first dose.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 876 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
RP2D (Phase 1) | Screening up to study completion, an average of 1 year.
AE (Phase 1) | Screening up to study completion, an average of 1 year.
Objective response rate (ORR) (Phase 2) | Screening up to study completion, an average of 1 year.

SECONDARY OUTCOMES:
Objective response rate (ORR) (Phase 1) | Screening up to study completion, an average of 1 year.
Disease control rate (DCR) (Phase 1) | Screening up to study completion, an average of 1 year.
Duration of response (DoR) (Phase 1) | Screening up to study completion, an average of 1 year.
Progression-free survival (PFS) (Phase 1) | Screening up to study completion, an average of 1 year.
Overall survival (OS) (Phase 1) | Screening up to study completion, an average of 1 year.
Drug Resistant Antibody (ADA) (Phase 1) | Screening up to study completion, an average of 1 year.
Blood concentration of SHR-1826 (Phase 1) | Screening up to study completion, an average of 1 year.
Blood concentration of free toxin SHR169265 (Phase 1) | Screening up to study completion, an average of 1 year.
Disease control rate (DCR) (Phase 2) | Screening up to study completion, an average of 1 year.
Duration of response (DoR) (Phase 2) | Screening up to study completion, an average of 1 year.
Progression-free survival (PFS) (Phase 2) | Screening up to study completion, an average of 1 year.
Overall survival (OS) (Phase 2) | Screening up to study completion, an average of 1 year.
AE (Phase 2) | Screening up to study completion, an average of 1 year.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen university cancer center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided